CLINICAL TRIAL: NCT01908751
Title: Fixation Using Alternative Implants for the Treatment of Hip Fractures (FAITH-2): A Multi-Centre 2x2 Factorial Randomized Trial Comparing Sliding Hip Screws Versus Cancellous Screws AND Vitamin D Versus Placebo on Patient Important Outcomes and Quality of Life in the Treatment of Young Adult (18-60) Femoral Neck Fractures
Brief Title: Fixation Using Alternative Implants for the Treatment of Hip Fractures (FAITH-2)
Acronym: FAITH-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Continuing beyond the pilot phase of the trial was deemed unfeasible
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster Surgical Associates (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Mohit Bhandari, Study Investigator, McMaster University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAITH-2
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Results first posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sliding Hip Screw and Vitamin D supplementation (Experimental): Participants allocated to the vitamin D Group will be given a six-month supply of vitamin D3 supplementation. Participants in the vitamin D Group will receive a bottle of 2,000 International Units (IU) vitamin D3 drops (Ddrops®, Ddrops Company). Participants will be instructed to take two drops daily for six months, for a total daily dose of 4,000 IU.
  Interventions: Procedure: Sliding Hip Screw; Drug: Vitamin D
- Sliding Hip Screw and Vitamin D placebo (Experimental): Participants in the placebo group will receive an identical bottle of placebo drops with no active ingredient. Similarly, they will be instructed to take two drops daily for six months. The placebo supplement is also manufactured by the Ddrops Company.
  Interventions: Procedure: Sliding Hip Screw; Drug: Vitamin D Placebo
- Cancellous Screws and Vitamin D supplementation (Experimental): Participants allocated to the vitamin D Group will be given a six-month supply of vitamin D3 supplementation. Participants in the vitamin D Group will receive a bottle of 2,000 International Units (IU) vitamin D3 drops (Ddrops®, Ddrops Company). Participants will be instructed to take two drops daily for six months, for a total daily dose of 4,000 IU.
  Interventions: Procedure: Cancellous Screws; Drug: Vitamin D
- Cancellous Screws and Vitamin D placebo (Experimental): Participants in the placebo group will receive an identical bottle of placebo drops with no active ingredient. Similarly, they will be instructed to take two drops daily for six months. The placebo supplement is also manufactured by the Ddrops Company.
  Interventions: Procedure: Cancellous Screws; Drug: Vitamin D Placebo

INTERVENTIONS:
Procedure: Sliding Hip Screw
  Arms: Sliding Hip Screw and Vitamin D placebo; Sliding Hip Screw and Vitamin D supplementation
Procedure: Cancellous Screws
  Arms: Cancellous Screws and Vitamin D placebo; Cancellous Screws and Vitamin D supplementation
Drug: Vitamin D
  Arms: Cancellous Screws and Vitamin D supplementation; Sliding Hip Screw and Vitamin D supplementation
Drug: Vitamin D Placebo
  Arms: Cancellous Screws and Vitamin D placebo; Sliding Hip Screw and Vitamin D placebo

SUMMARY:
The purpose of this study is to determine the impact of surgical fixation (cancellous screws versus sliding hip screws) and biologic intervention (Vitamin D versus placebo) on patient important outcomes.

DETAILED DESCRIPTION:
Femoral neck fractures are a type of hip fracture associated with high complication rates and poor functional outcomes. It is estimated that over 300,000 hip fractures occur in patients under age 50 annually. Hip fractures in younger aged patients are particularly devastating with profound impairments of quality of life and function. Virtually all patients require surgical repair of their fractures and unlike elderly hip fractures, failure of surgery offers few options for salvage. Arthroplasty is a successful treatment for elderly patients; however, a hip replacement is not a viable option for younger patients because of their higher functional demands for work and recreational activities that are not tolerated by joint replacements.

There is more than one way to perform internal fixation for femoral neck fractures. Cancellous screws have traditionally been the preferred internal fixation implant for femoral neck fractures. Multiple screws (2 or more) are used during fixation, and advocates of this implant promote the construct's superior torsional stability, limited disruption of femoral head blood supply, minimally invasive insertion, and retention of more viable bone than the larger sliding hip screw (SHS). On the other hand, sliding hip screws have been gaining popularity and there is evidence to suggest that SHS provide greater fracture stability and may reduce patient complications. It is currently unknown which method of internal fixation provides the best outcomes for patients.

Femoral neck fracture treatment is further complicated by vitamin D insufficiency in as many as 8 of 10 trauma patients. Vitamin D plays an important role in musculoskeletal health and bone quality because it regulates serum calcium homeostasis. Laboratory research and human clinical studies suggest important associations between vitamin D, musculoskeletal health, and improved fracture healing. Experimental animal studies have demonstrated the concentration of vitamin D metabolites are higher at a fracture callus compared to the uninjured contralateral bone, vitamin D supplementation leads to decreased time to fracture union and increased callus vascularity, and vitamin D increases mechanical bone strength compared to controls. Clinical studies have also demonstrated that vitamin D supplementation increases the callus volume of proximal humerus fractures, increases the number and diameter of type II muscle fibres, and can improve wound healing, however, the effects of vitamin D supplementation in you patients with femoral neck fractures are unknown.

Using a 2x2 factorial design, participant will be randomly allocated to one of four treatment arms. Participants allocated to the cancellous screw group will receive multiple threaded screws (with a minimum of 3 screws and a minimum diameter of 6.5 mm) and those allocated to the sliding hip screw group will receive a single larger diameter partially threaded screw affixed to the proximal femur with a sideplate using a minimum of 2 screws for fixation. Participants allocated to the vitamin D Group will receive a bottle of 2,000 International Units (IU) vitamin D3 drops. Participants will be instructed to take two drops daily for six months, for a total daily dose of 4,000 IU. Participants in the placebo group will receive an identical bottle of placebo drops with no active ingredient. Similarly, they will be instructed to take two drops daily for six months. All vitamin D3 supplement and placebo bottles will be labeled in a blinded manner according to Health Canada and Good Manufacturing Practice.

Participation in this study will last 12 months. In-person participant follow-up visits will occur at enrollment (baseline), post-surgery, 6 weeks, 3 months, 6 months, 9 months, and 12 months post-surgery. Data for all outcomes and radiographs will be collected at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria

1. Adult men or women ages 18 to 60 years.
2. Fracture of the femoral neck.
3. Fracture amenable to both surgical treatments (SHS and cancellous screws).
4. Operative treatment within 7 days of injury.
5. Provision of informed consent by patient or substitute decision maker.

Exclusion Criteria

1. Patients with previously diagnosed osteoporosis.
2. Fracture-dislocation of the femoral neck and hip joint.
3. Planned antegrade nailing of an ipsilateral femoral shaft fracture (if present).
4. Current infection around the hip (i.e. soft tissue or bone).
5. Stress fracture of the femoral neck.
6. Pathologic fractures secondary to neoplasm or other bone lesion.
7. Patients with known or likely undiagnosed disorders of bone metabolism such as Paget's disease, osteomalacia, osteopetrosis, osteogenesis imperfect, etc.
8. Patients with hyperhomocysteinemia.
9. Patient has an allergy to vitamin D or another contraindication to being prescribed vitamin D.
10. Patient is currently taking an over counter drug and/or food supplement that contains vitamin D and is unable or unwilling to discontinue its use for this study.
11. Likely problems, in the judgment of the attending surgeon, with maintaining follow up (e.g. patients with no fixed address, plans to move out of town). This may include patients with severe mental disorders and drug addictions without adequate support.
12. Pregnancy.
13. Patient is incarcerated.
14. Patient is not expected to survive injuries.
15. The attending surgeon believes the patient should be excluded because they are involved in a conflicting clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2014-09; Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Slobogean, MD, Principal Investigator — University of Maryland, College Park; Mohit Bhandari, MD, Principal Investigator — McMaster University; Sheila Sprague, PhD, Study Director — McMaster University (Role: Research Methodologist)
Locations (20):
- United States (10):
  - The Center for Orthopedic Research and Education (CORE) Institute, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Indiana University (IU Health Methodist Hospital), Indianapolis, Indiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Hennepin Healthcare System, Minneapolis, Minnesota
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Inova Health Care Services, Falls Church, Virginia
  - West Virginia University, Morgantown, West Virginia
- Alfred Health, Melbourne, Victoria, Australia
- Canada (9):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - University of British Columbia & Vancouver Costal Health Authority, Vancouver, British Columbia
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Memorial University, St. John's, Newfoundland and Labrador
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Background] Baitner AC, Maurer SG, Hickey DG, Jazrawi LM, Kummer FJ, Jamal J, Goldman S, Koval KJ. Vertical shear fractures of the femoral neck. A biomechanical study. Clin Orthop Relat Res. 1999 Oct;(367):300-5. PMID 10546628
- [Background] Bee CR, Sheerin DV, Wuest TK, Fitzpatrick DC. Serum vitamin D levels in orthopaedic trauma patients living in the northwestern United States. J Orthop Trauma. 2013 May;27(5):e103-6. doi: 10.1097/BOT.0b013e31825cf8fb. PMID 22576645
- [Background] Bhandari M, Devereaux PJ, Swiontkowski MF, Tornetta P 3rd, Obremskey W, Koval KJ, Nork S, Sprague S, Schemitsch EH, Guyatt GH. Internal fixation compared with arthroplasty for displaced fractures of the femoral neck. A meta-analysis. J Bone Joint Surg Am. 2003 Sep;85(9):1673-81. doi: 10.2106/00004623-200309000-00004. PMID 12954824
- [Background] Bhandari M, Tornetta P 3rd, Hanson B, Swiontkowski MF. Optimal internal fixation for femoral neck fractures: multiple screws or sliding hip screws? J Orthop Trauma. 2009 Jul;23(6):403-7. doi: 10.1097/BOT.0b013e318176191f. PMID 19550225
- [Background] Chen Z, Wang G, Lin J, Yang T, Fang Y, Liu L, Zhang H. [Efficacy comparison between dynamic hip screw combined with anti-rotation screw and cannulated screw in treating femoral neck fractures]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2011 Jan;25(1):26-9. Chinese. PMID 21351604
- [Background] Damany DS, Parker MJ, Chojnowski A. Complications after intracapsular hip fractures in young adults. A meta-analysis of 18 published studies involving 564 fractures. Injury. 2005 Jan;36(1):131-41. doi: 10.1016/j.injury.2004.05.023. PMID 15589931
- [Background] Doetsch AM, Faber J, Lynnerup N, Watjen I, Bliddal H, Danneskiold-Samsoe B. The effect of calcium and vitamin D3 supplementation on the healing of the proximal humerus fracture: a randomized placebo-controlled study. Calcif Tissue Int. 2004 Sep;75(3):183-8. doi: 10.1007/s00223-004-0167-0. PMID 15386160
- [Background] Hamilton B. Vitamin D and human skeletal muscle. Scand J Med Sci Sports. 2010 Apr;20(2):182-90. doi: 10.1111/j.1600-0838.2009.01016.x. Epub 2009 Oct 5. PMID 19807897
- [Background] Johansson A, Stromqvist B, Bauer G, Hansson LI, Pettersson H. Improved operations for femoral neck fracture. A radiographic evaluation. Acta Orthop Scand. 1986 Dec;57(6):505-9. doi: 10.3109/17453678609014779. PMID 3577716
- [Background] Langlois K, Greene-Finestone L, Little J, Hidiroglou N, Whiting S. Vitamin D status of Canadians as measured in the 2007 to 2009 Canadian Health Measures Survey. Health Rep. 2010 Mar;21(1):47-55. PMID 20426226
- [Background] Lappe J, Cullen D, Haynatzki G, Recker R, Ahlf R, Thompson K. Calcium and vitamin d supplementation decreases incidence of stress fractures in female navy recruits. J Bone Miner Res. 2008 May;23(5):741-9. doi: 10.1359/jbmr.080102. PMID 18433305
- [Background] Lidor C, Dekel S, Hallel T, Edelstein S. Levels of active metabolites of vitamin D3 in the callus of fracture repair in chicks. J Bone Joint Surg Br. 1987 Jan;69(1):132-6. doi: 10.1302/0301-620X.69B1.3029136.
- [Background] Linde F, Andersen E, Hvass I, Madsen F, Pallesen R. Avascular femoral head necrosis following fracture fixation. Injury. 1986 May;17(3):159-63. doi: 10.1016/0020-1383(86)90322-0. PMID 3818052
- [Background] Lindequist S. Cortical screw support in femoral neck fractures. A radiographic analysis of 87 fractures with a new mensuration technique. Acta Orthop Scand. 1993 Jun;64(3):289-93. doi: 10.3109/17453679308993627. PMID 8322583
- [Background] Malchau H, Herberts P, Eisler T, Garellick G, Soderman P. The Swedish Total Hip Replacement Register. J Bone Joint Surg Am. 2002;84-A Suppl 2:2-20. doi: 10.2106/00004623-200200002-00002. No abstract available. PMID 12479335
- [Background] Omeroglu H, Ates Y, Akkus O, Korkusuz F, Bicimoglu A, Akkas N. Biomechanical analysis of the effects of single high-dose vitamin D3 on fracture healing in a healthy rabbit model. Arch Orthop Trauma Surg. 1997;116(5):271-4. doi: 10.1007/BF00390051. PMID 9177802
- [Background] Omeroglu S, Erdogan D, Omeroglu H. Effects of single high-dose vitamin D3 on fracture healing. An ultrastructural study in healthy guinea pigs. Arch Orthop Trauma Surg. 1997;116(1-2):37-40. PMID 9006763
- [Background] Patil S, Garbuz DS, Greidanus NV, Masri BA, Duncan CP. Quality of life outcomes in revision vs primary total hip arthroplasty: a prospective cohort study. J Arthroplasty. 2008 Jun;23(4):550-3. doi: 10.1016/j.arth.2007.04.035. Epub 2007 Oct 23. PMID 18514873
- [Background] Sakalli H, Arslan D, Yucel AE. The effect of oral and parenteral vitamin D supplementation in the elderly: a prospective, double-blinded, randomized, placebo-controlled study. Rheumatol Int. 2012 Aug;32(8):2279-83. doi: 10.1007/s00296-011-1943-6. Epub 2011 May 10. PMID 21556746
- [Background] Swiontkowski MF, Harrington RM, Keller TS, Van Patten PK. Torsion and bending analysis of internal fixation techniques for femoral neck fractures: the role of implant design and bone density. J Orthop Res. 1987;5(3):433-44. doi: 10.1002/jor.1100050316. PMID 3625366
- [Derived] FAITH-2 Investigators; Slobogean GP, Sprague S, Bzovsky S, Heels-Ansdell D, Thabane L, Scott T, Bhandari M. Fixation using alternative implants for the treatment of hip fractures (FAITH-2): design and rationale for a pilot multi-centre 2 x 2 factorial randomized controlled trial in young femoral neck fracture patients. Pilot Feasibility Stud. 2019 May 28;5:70. doi: 10.1186/s40814-019-0458-x. eCollection 2019. PMID 31161044

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 91 patients were enrolled into the FAITH-2 pilot trial. Five of these enrolments were subsequently determined to be ineligible (not between the ages of 18-60 years, pathological fracture, no femoral neck fracture, did not provide informed consent (2 patients)). Therefore, 86 participants were included in the analysis.
Groups:
- Sliding Hip Screw + Vitamin D Supplementation: Participants allocated to this group received a single larger diameter partially threaded screw affixed to the proximal femur with a side plate and were given a six-month supply of vitamin D3 supplementation. Participants in the vitamin D Group received a bottle of 2,000 International Units (IU) vitamin D3 drops (Ddrops®, Ddrops Company). Participants were instructed to take two drops daily for six months, for a total daily dose of 4,000 IU.
- Cancellous Screws + Vitamin D Supplementation: Participants allocated to this group received multiple cancellous screws with a minimum diameter of 6.5 mm and were given a six-month supply of vitamin D3 supplementation. Participants in the vitamin D Group received a bottle of 2,000 International Units (IU) vitamin D3 drops (Ddrops®, Ddrops Company). Participants were instructed to take two drops daily for six months, for a total daily dose of 4,000 IU.
- Sliding Hip Screw + Vitamin D Placebo: Participants allocated to this group received a single larger diameter partially threaded screw affixed to the proximal femur with a side plate and were given an identical bottle of placebo drops with no active ingredient. Similarly, they were instructed to take two drops daily for six months. The placebo supplement was also manufactured by the Ddrops Company.
- Cancellous Screws + Vitamin D Placebo: Participants allocated to this group received multiple cancellous screws with a minimum diameter of 6.5 mm and were given an identical bottle of placebo drops with no active ingredient. Similarly, they were instructed to take two drops daily for six months. The placebo supplement was also manufactured by the Ddrops Company.
Period: Overall Study
Arm/Group | Sliding Hip Screw + Vitamin D Supplementation | Cancellous Screws + Vitamin D Supplementation | Sliding Hip Screw + Vitamin D Placebo | Cancellous Screws + Vitamin D Placebo
Started | 22 | 23 | 21 | 20
Completed | 17 | 18 | 16 | 16
Not Completed | 5 | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sliding Hip Screw + Vitamin D Supplementation | Cancellous Screws + Vitamin D Supplementation | Sliding Hip Screw + Vitamin D Placebo | Cancellous Screws + Vitamin D Placebo | Total
Number analyzed (Participants) | 22 | 23 | 21 | 20 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (11.2) | 40.3 (13.0) | 45.2 (11.5) | 37.9 (13.7) | 41.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 8 | 3 | 23
  Male | 17 | 16 | 13 | 17 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indigenous | 0 | 0 | 1 | 0 | 1
  South Asian | 1 | 0 | 0 | 1 | 2
  Southeast Asian (Filipino) | 0 | 0 | 1 | 0 | 1
  Hispanic/Latino | 1 | 0 | 0 | 1 | 2
  White | 14 | 19 | 18 | 17 | 68
  Black | 4 | 3 | 1 | 1 | 9
  Mixed (Black & White) | 1 | 0 | 0 | 0 | 1
  Middle Eastern | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 7 | 7 | 7 | 28
  United States | 15 | 16 | 14 | 13 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Patient Important Outcomes
Description: A participant met the primary clinical endpoint if they experienced one or more of the four outcomes:
  1. Re-operation: any unplanned surgery related to the treatment of the femoral neck fracture;
  2. Femoral head osteonecrosis: any evidence of osteonecrosis on any follow-up medical imaging study (i.e., radiographs, magnetic resonance imaging (MRI), or other advanced imaging study);
  3. Severe femoral neck malunion: fracture healing with femoral neck shortening of >10 mm in any plane on follow-up x-rays; or
  4. Nonunion: failure of the fracture to progress towards healing defined as a Radiographic Union Score for Hip (RUSH) score below a pre-determined threshold specific for nonunion at 6 months or greater post-injury.
Time Frame: 12 months post-surgery
Population: 91 patients were randomized into the FAITH-2 pilot trial. 86 patients were deemed eligible and included in the analyses. Of the 86 participants, 43 were allocated to receive a sliding hip screw and 43 were allocated to receive CS. Regarding supplementation treatment, 45 were allocated to receive vitamin D, and 41 were allocated to receive placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Sliding Hip Screw: Participants allocated to the Sliding Hip Screw group received a single larger diameter partially threaded screw affixed to the proximal femur with a side plate.
- Cancellous Screws: Participants allocated to the Cancellous Screws group received multiple cancellous screws with a minimum diameter of 6.5 mm.
- Vitamin D Supplementation: Participants allocated to the vitamin D Group were given a six-month supply of vitamin D3 supplementation. Participants in the vitamin D Group received a bottle of 2,000 International Units (IU) vitamin D3 drops (Ddrops®, Ddrops Company). Participants were instructed to take two drops daily for six months, for a total daily dose of 4,000 IU.
- Vitamin D Placebo: Participants in the placebo group received an identical bottle of placebo drops with no active ingredient. Similarly, they were instructed to take two drops daily for six months. The placebo supplement was also manufactured by the Ddrops Company.
Arm/Group | Sliding Hip Screw | Cancellous Screws | Vitamin D Supplementation | Vitamin D Placebo
Number analyzed (Participants) | 43 | 43 | 45 | 41
Participants
  Primary Clinical Endpoint | 11 | 13 | 11 | 13
  Re-operation | 9 | 6 | 7 | 8
  Femoral head osteonecrosis | 2 | 7 | 5 | 4
  Severe femoral neck malunion | 2 | 6 | 5 | 3
  Nonunion | 4 | 3 | 4 | 3

2. Secondary Outcome: Number of Participants With Non-Operatively-Treated Fracture Healing Complications
Description: Fracture healing complications treated non-operatively are presented in this table and included wound healing problems, infection (superficial and deep), hardware failure, hardware breakage, painful hardware, and peri-prosthetic fracture.
Time Frame: 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Sliding Hip Screw | Cancellous Screws | Vitamin D Supplementation | Vitamin D Placebo
Number analyzed (Participants) | 43 | 43 | 45 | 41
Participants | 0 | 1 | 0 | 0

3. Secondary Outcome: Short Form-12 (SF-12) Physical Composite Scale (PCS)
Description: The SF-12 is a 12-item questionnaire that measures self-reported quality of life through an 8-domain profile of functional health and well-being, physical and mental health summary measures and a preference-based health utility index. Scores range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Pre-fracture, 6 weeks, 3 months, 6 months, 9 months, 12 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sliding Hip Screw | Cancellous Screws | Vitamin D Supplementation | Vitamin D Placebo
Number analyzed (Participants) | 43 | 43 | 45 | 41
scores on a scale
  Pre-fracture | 50.5 (10.4) | 53.7 (7.1) | 53.5 (7.1) | 50.8 (10.5)
  6 Weeks | 29.9 (8.5) | 29.3 (10.2) | 29.7 (9.6) | 29.4 (9.2)
  3 Months | 36.2 (11.2) | 36.7 (10.7) | 37.2 (12.0) | 35.7 (9.5)
  6 Months | 36.9 (11.5) | 43.4 (13.0) | 41.4 (12.9) | 38.8 (12.4)
  9 Months | 38.3 (12.8) | 45.0 (13.2) | 41.8 (14.0) | 42.4 (12.5)
  12 Months | 42.2 (12.4) | 45.0 (11.6) | 44.5 (10.9) | 42.6 (13.3)

4. Secondary Outcome: Short Form-12 (SF-12) Mental Health Composite Scale (MCS)
Description: The SF-12 is a 12-item questionnaire that measures self-reported quali... If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome. Scores range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Pre-fracture, 6 weeks, 3 months, 6 months, 9 months, 12 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sliding Hip Screw | Cancellous Screws | Vitamin D Supplementation | Vitamin D Placebo
Number analyzed (Participants) | 43 | 43 | 45 | 41
scores on a scale
  Pre-fracture | 55.6 (8.1) | 53.1 (8.3) | 54.3 (7.6) | 54.2 (9.0)
  6 Weeks | 52.0 (11.5) | 53.9 (9.9) | 53.0 (9.8) | 52.9 (11.8)
  3 Months | 50.5 (13.2) | 54.3 (10.1) | 54.4 (10.3) | 50.1 (13.2)
  6 Months | 55.0 (9.9) | 54.2 (8.6) | 52.9 (8.2) | 57.0 (10.2)
  9 Months | 54.0 (9.7) | 54.0 (9.9) | 53.8 (10.0) | 54.3 (9.5)
  12 Months | 52.9 (9.8) | 53.3 (9.2) | 52.4 (9.3) | 53.9 (9.6)

5. Secondary Outcome: Hip Outcome Score (HOS) Activities of Daily Living Scale
Description: The HOS measures self-reported functional status through 28 items and two sub-scales that pertain to activities of daily living (ADLs) or higher level activities such as those necessary to participate in sports. Scores for each subscale range from 0 (least function) to 100 (most function).
Time Frame: Pre-fracture, 6 weeks, 3 months, 6 months, 9 months, 12 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sliding Hip Screw | Cancellous Screws | Vitamin D Supplementation | Vitamin D Placebo
Number analyzed (Participants) | 43 | 43 | 45 | 41
scores on a scale
  Pre-fracture | 89.2 (20.4) | 95.4 (14.8) | 93.1 (18.3) | 91.5 (17.7)
  6 Weeks | 39.1 (19.5) | 36.1 (23.1) | 38.1 (23.1) | 37.1 (19.0)
  3 Months | 56.8 (24.1) | 59.3 (25.5) | 56.7 (25.4) | 59.8 (23.7)
  6 Months | 64.5 (24.4) | 74.4 (23.1) | 69.7 (23.8) | 69.6 (25.0)
  9 Months | 69.0 (21.1) | 79.6 (22.4) | 75.1 (23.2) | 74.7 (21.4)
  12 Months | 73.0 (22.7) | 79.4 (22.7) | 76.6 (21.5) | 76.2 (23.5)

6. Secondary Outcome: Hip Outcome Score (HOS) Sports Scale
Description: as for outcome 5
Time Frame: Pre-fracture, 6 weeks, 3 months, 6 months, 9 months, 12 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sliding Hip Screw | Cancellous Screws | Vitamin D Supplementation | Vitamin D Placebo
Number analyzed (Participants) | 43 | 43 | 45 | 41
scores on a scale
  Pre-fracture | 78.5 (33.5) | 86.9 (25.9) | 88.6 (25.5) | 76.4 (33.3)
  6 Weeks | 9.3 (14.9) | 8.0 (13.4) | 8.0 (13.7) | 9.4 (14.7)
  3 Months | 20.8 (22.9) | 21.4 (25.1) | 20.1 (23.8) | 22.2 (23.9)
  6 Months | 33.0 (31.0) | 45.1 (28.7) | 38.1 (30.7) | 41.0 (29.5)
  9 Months | 42.8 (33.9) | 54.8 (28.7) | 52.4 (33.0) | 45.6 (29.2)
  12 Months | 47.5 (31.0) | 57.3 (31.4) | 52.4 (33.4) | 53.1 (29.6)

7. Secondary Outcome: Radiographic Fracture Healing
Description: The date of healing will be determined by the Central Adjudication Committee (CAC). They will consider a fracture as healed when there is obliteration of the fracture line by newly formed bone along the cortices and within the trabecular bone on anterior-posterior and lateral radiographs.
Time Frame: up to 12 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sliding Hip Screw | Cancellous Screws | Vitamin D Supplementation | Vitamin D Placebo
Number analyzed (Participants) | 43 | 43 | 45 | 41
days | 224.0 (131.5) | 236.7 (136.7) | 210.4 (121.0) | 252.3 (144.2)

ADVERSE EVENTS:
Time Frame: 12 months
Description: An AE is any symptom, sign, illness, or experience that develops or worsens in severity during the course of this study. AEs are classified as serious or non-serious. A SAE is any AE that is any of the following:
  * Fatal
  * Life threatening
  * Requires or prolongs hospital stay
  * Results in persistent or significant disability or incapacity
  * A congenital anomaly or birth defect
  * An important medical event
Arm/Group | Sliding Hip Screw + Vitamin D Supplementation | Cancellous Screws + Vitamin D Supplementation | Sliding Hip Screw + Vitamin D Placebo | Cancellous Screws + Vitamin D Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 5/22 | 6/23 | 9/21 | 5/20
Other Adverse Events (participants affected / at risk) | 2/22 | 3/23 | 3/21 | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sliding Hip Screw + Vitamin D Supplementation (N=22) | Cancellous Screws + Vitamin D Supplementation (N=23) | Sliding Hip Screw + Vitamin D Placebo (N=21) | Cancellous Screws + Vitamin D Placebo (N=20)
Aortic valve replacement due to intravalvular prosthetic regurgitation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Painful Hardware or Hardware Failure/Breakage (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (5) | 1 (1)
Nonunion (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Osteonecrosis, symptomatic (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Post-traumatic femoral acetabular impingement & hip range of motion restrictions (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (deep) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sliding Hip Screw + Vitamin D Supplementation (N=22) | Cancellous Screws + Vitamin D Supplementation (N=23) | Sliding Hip Screw + Vitamin D Placebo (N=21) | Cancellous Screws + Vitamin D Placebo (N=20)
Delayed Union (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteonecrosis, asymptomatic (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Accident/Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash/Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Meniscal tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT01908751/Prot_SAP_000.pdf